CLINICAL TRIAL: NCT05795478
Title: Effects of Oxycodone Combined With Pregabalin on Chronic Postsurgical Pain in Spinal Surgery: a Randomized Control, Double-blinded, Factorial Design Trial
Brief Title: Effects of Oxycodone Combined With Pregabalin on Chronic Postsurgical Pain in Spinal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Director of Anesthesiology Department, Beijing Tiantan Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: sunQKT6660
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Chronic Post Operative Pain; Oxycodone; Pregabalin; Postoperative Complications
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Oxycodone; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combined group (Experimental): Oxycodone+Pregabalin
  Interventions: Drug: Oxycodone and Pregabalin
- Oxycodone group (Other): Oxycodone+placebo capsules
  Interventions: Drug: Oxycodone and placebo capsules
- Pregabalin group (Other): NS+Pregabalin
  Interventions: Drug: Pregabalin and NS
- Control group (Placebo Comparator): NS+placebo capsules
  Interventions: Drug: placebo capsules and NS

INTERVENTIONS:
Drug: Oxycodone and Pregabalin — Oxycodone: 150mg PCIA during 3 days postoperatively Pregabalin: 150mg preoperatvely, 75mg BID for POD1~7,75mg QD for POD8~14
  Arms: Combined group
Drug: Oxycodone and placebo capsules — Oxycodone: 150mg PCIA for 3 days postoperatively placebo capsules: same numbers as pregabalin at each time point
  Arms: Oxycodone group
Drug: Pregabalin and NS — Pregabalin: 150mg preoperatively, 75mg BID for POD1~7,75mg QD for POD8~14 NS: Equal volume NS for 3 days postoperatively
  Arms: Pregabalin group
Drug: placebo capsules and NS — placebo capsules: same numbers as pregabalin at each time point NS: Equal volume NS for 3 days postoperatively
  Arms: Control group

SUMMARY:
Chronic postoperative pain is one of the common perioperative complications, which seriously affects the prognosis of patients. Currently, no specific perioperative pain management strategy has been found to be effective in preventing and treating chronic postoperative pain in patients undergoing spinal surgery. At present, oxycodone has been widely recognized in different surgical populations for the control of acute postoperative pain, but its contribution to chronic postoperative pain remains unknown. Meanwhile, whether pregabalin can reduce the occurrence of chronic postoperative pain remains controversial, and whether the combination of the two drugs can control the occurrence of chronic postoperative pain in a more comprehensive way remains unknown. Therefore, we intend to conduct this randomized-controlled, factorial design study to determine the efficacy and safety of oxycodone combined with pregabalin in the treatment of chronic postoperative pain in patients undergoing spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective spinal surgery
* Ages equal to or more than 18 years old
* ASA I-III
* Signed informed consent

Exclusion Criteria:

* Previous allergic history to gabapentinoids or oxycodone;
* Patients with aphasia or inability to cooperate with scales assessments;
* Patients with a diagnosed history of psychiatric disorder;
* Known severe insufficiency of vitals(such as heart failure/renal dysfunction/hepatic failure);
* Patients treated with gabapentin/pregabalin in the last three months;
* History of drug abuse;
* Body Mass Index more than 35 kg/㎡;
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of CPSP | 3 months after surgery
  The incidence of chronic postsurgical pain, the CPSP was defined as an NRS score >3 (0~10).

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph D., Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China